CLINICAL TRIAL: NCT05911945
Title: Failed Insertion of Ureteral Access Sheath During Flexible Ureterorenoscopy: A Randomized Controlled Trial Comparing Second Session Flexible Ureterorenoscopy or Same Session Mini Percutaneous Nephrolithotomy
Brief Title: Failed Insertion of Ureteral Access Sheath During Flexible Ureterorenoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ufuk Çağlar, M.D, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 256040791
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Kidney Calculi
Keywords: kidney calculi; percutaneous nephrolithotomy; retrograde intrarenal surgery; quality of life
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Ureterorenoscopy (Active Comparator): Underwent a JJ stent insertion and underwent f-URS 4-6 weeks later (Group 1).
  Interventions: Procedure: Flexible Ureterorenoscopy
- Mini Percutaneous Nephrolithotomy (Active Comparator): Underwent mPNL operation in the same session after prone positioning (Group 2).
  Interventions: Procedure: Mini Percutaneous Nephrolithotomy

INTERVENTIONS:
Procedure: Flexible Ureterorenoscopy — A guidewire was placed in the ureter in the lithotomy position. Ureterorenoscopy was performed with an 8 Fr ureterorenoscope for active dilatation. An 11 - 13 Fr or 9.5 / 11.5 Fr UAS was attempted to be placed under fluoroscopy by the surgeon of the procedure. In cases where the UAS could not inserted, a 26 cm, 4.8 Fr JJ stent was placed under fluoroscopy and the procedure was terminated. Patients underwent a second f-URS session, 4 - 6 weeks later. After the JJ stent was removed, an 11 - 13 Fr UAS was placed in the ureter. Digital flexible ureterorenoscope was used as the flexible ureteroscope. Stone fragmentation was performed in dusting mode using a Ho:YAG laser with a 272 µ probe. After fragmentation, a 26 cm 4.8 Fr JJ stent was inserted into the ureter. The JJ stent was removed at 4 - 6 weeks postoperatively.
  Arms: Flexible Ureterorenoscopy
Procedure: Mini Percutaneous Nephrolithotomy — A guidewire was placed in the ureter in the lithotomy position. Ureterorenoscopy was performed with an 8 Fr ureterorenoscope for active dilatation. An 11 - 13 Fr or 9.5 / 11.5 Fr UAS was attempted to be placed under fluoroscopy by the surgeon of the procedure. In cases where the UAS could not inserted, patients were positioned in prone position and access was performed to the appropriate calyx with an 18-gauge percutaneous access needle using the triangulation technique accompanied by fluoroscopy, in the same session. After the guidewire was introduced into the pelvicalyceal system, sequential dilatation was applied with Amplatz dilatators, and a 21 Fr metallic sheath was placed. Stones were fragmented with a yttrium-aluminum-garnet (Ho:YAG) Laser lithotripter. At the end of the procedure, a 14 Fr nephrostomy catheter was placed in according to the residual stone, hemorrhage, and perforation status. In other cases, the procedure was concluded as totally tubeless.
  Arms: Mini Percutaneous Nephrolithotomy

SUMMARY:
Percutaneous nephrolithotomy (PNL) is the gold standard recommended treatment technique for kidney stones larger than 20 mm. For kidney stones between 10 - 20 mm, both shock wave lithotripsy (SWL) or flexible ureterorenoscopy (f-URS) are recommended as the first choice of treatment and PNL is recommended as the second. In patients who are planned to undergo f-URS, a ureteral access sheath (UAS) is placed in the ureter at the beginning of the operation in order to provide a better image, reduce intra-renal pressure, easier stone fragment retrieval and shorter operative time. In certain cases, such as ureteral stricture, kink or edema, the ureteral access sheath may not be able to successfully inserted into the ureter. At this stage, double-J (JJ) stent can be inserted into the ureter to create passive dilatation, and a second f-URS session can be scheduled a few weeks later. Another option is to perform PNL operation to the patient in the same session. In this randomized prospective study, we aimed to compare these two different surgical approaches in terms of patient comfort and surgical success in patients with kidney stones between 10 - 20 mm in which access sheath insertion was failed in the initial f-URS session.

DETAILED DESCRIPTION:
Patients with renal calculi between 1 - 2 cm in diameter who were admitted to a tertiary health institution were evaluated prospectively. Patients who were unsuitable for shock wave lithotripsy (SWL) treatment or who did not benefit from SWL sessions were included in the study. Randomization was performed using a random number table with a central computerized system. Before the procedure, the patients were asked to complete the Turkish language validated form of the Short Form - 36 (SF - 36) questionnaire.

A total of 48 patients in whom ureteral access sheath insertion has failed during initial flexible ureterorenoscopy (f-URS) session were randomly divided into 2 groups. Group 1 underwent a JJ stent insertion and procedure terminated, while group 2 underwent mini percutaneous nephrolithotomy (mPNL) operation in the same session after prone positioning. Group 1 underwent f-URS 4-6 weeks later. One month after the operation, stone-free status was evaluated with computed tomography (CT) and detection of residual fragments of any size was defined as failure. The patients were asked to fill out the SF-36 questionnaire one month after the last surgery. Operative and postoperative data, SF-36 results, success, and complications were compared between the groups. The operation time included the time from initiation of cystoscopy to removal of amplatz for the mPNL group. For the F-URS group, it was calculated as the sum of the times between cystoscopy and fluoroscopy control of the JJ stent in both sessions.

Surgical technique All surgeries were performed by the same team of experienced surgeons in with high expertise in endourology. A guidewire was placed in the ureter in the lithotomy position. Ureterorenoscopy was performed with an 8 Fr ureterorenoscope for active dilatation. An 11 - 13 Fr or 9.5 / 11.5 Fr UAS was attempted to be placed under fluoroscopy by the surgeon of the procedure. In cases where the UAS could not inserted, a 26 cm, 4.8 Fr JJ stent was placed under fluoroscopy in the f-URS group, and the procedure was terminated. In the mPNL group, same session mPNL procedure was performed.

After initial JJ stent placement, patients in group 1 underwent a second f-URS session, 4 - 6 weeks later. After the JJ stent was removed, an 11 - 13 Fr UAS was placed in the ureter. Digital flexible ureterorenoscope was used as the flexible ureteroscope. Stone fragmentation was performed in dusting mode using a Ho:YAG laser with a 272 µ probe. After fragmentation, a 26 cm 4.8 Fr JJ stent was inserted into the ureter. The JJ stent was removed at 4 - 6 weeks postoperatively.

For patients in group 2, after placing a 5 Fr ureteral open-ended catheter, patients were positioned in prone position and access was performed to the appropriate calyx with an 18-gauge percutaneous access needle using the triangulation technique accompanied by fluoroscopy, in the first session. After the guidewire was introduced into the pelvicalyceal system, sequential dilatation was applied with Amplatz dilatators, and a 21 Fr metallic sheath was placed. Stones were fragmented with a yttrium-aluminum-garnet (Ho:YAG) Laser lithotripter. At the end of the procedure, a 14 Fr nephrostomy catheter was placed in according to the residual stone, hemorrhage, and perforation status. In other cases, the procedure was concluded as totally tubeless. Postoperative routine intravenous analgesia was not applied to all patients.

Study sample size analysis was computed using the G*Power program (effect size 0.5, alfa error 0.05, power 0.80). Statistical analysis was performed with 'Statistical Package for the Social Sciences' (SPSS) 25 program. The normality assessment of the distribution of the data was analyzed with the Shapiro-Wilk test and Q - Q plot. For continuous covariates, normality and homogeneity of each variable were evaluated and Student's or Welch's t-test was performed. Mann - Whitney U test was used for skewed data. Quantitative data were presented as mean ± standard deviation or median (IQR) values. Chi-square test or Fisher exact test (where the 20% of expected cell counts were less than 5) was used to compare qualitative data. The normality of the differences in SF - 36 data before and after the procedure was evaluated with the Skewness test and Q - Q plot. Paired-sample t - test was used to compare SF - 36 data before and after the procedure. The data were analyzed at 95% confidence level and the values with P < .05 were noted statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal calculi between 1 - 2 cm in diameter
* Patients who were unsuitable for SWL treatment or who did not benefit from SWL sessions

Exclusion Criteria:

* Patients with kidney anomalies, (malrotated and horseshoe kidneys, kidneys with duplicated systems)
* Pregnant patients
* Patients younger than 18 years of age
* Patients who did not consent for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Short Form-36 parameters | Before surgery - 1 month after surgery
  In order to evaluate the quality of life of the patients, pre- and postoperative SF-36 form values will be compared.

SECONDARY OUTCOMES:
The success of the surgery | Before surgery - 1 month after surgery
  Stone-free rates of the patients will be evaluated by computed tomography after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akbulut, Assoc. Prof, Study Director — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang K, Zhang P, Xu B, Luo G, Hu J, Zhu J, Sun F. Percutaneous Nephrolithotomy vs. Retrograde Intrarenal Surgery for Renal Stones Larger than 2cm in Patients with a Solitary Kidney: A Systematic Review and a Meta-Analysis. Urol J. 2020 Jul 28;17(5):442-448. doi: 10.22037/uj.v16i7.5609. PMID 32748387
- [Background] Bensalah K, Tuncel A, Gupta A, Raman JD, Pearle MS, Lotan Y. Determinants of quality of life for patients with kidney stones. J Urol. 2008 Jun;179(6):2238-43; discussion 2243. doi: 10.1016/j.juro.2008.01.116. Epub 2008 Apr 18. PMID 18423704
- [Background] Perez-Fentes DA, Gude F, Blanco B, Freire CG. Percutaneous nephrolithotomy: short- and long-term effects on health-related quality of life. J Endourol. 2015 Jan;29(1):13-7. doi: 10.1089/end.2014.0081. PMID 24708396